CLINICAL TRIAL: NCT02160704
Title: PHASE 2b RANDOMIZED, PARALLEL, DOUBLE-BLIND, PLACEBO-CONTROLLED EXPLORATORY STUDY TO EVALUATE THE EFFICACY OF ANDROXAL IN IDIOPATHIC MALE INFERTILITY (PROTOCOL #01-14-40-08)
Brief Title: Androxal in Male Infertility
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Difficult eligibility and lack of funding
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Larry I. Lipshultz, Professor of Urology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-33673
Record Dates: First submitted 2014-06-05; First posted 2014-06-11 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Infertility
Keywords: Sperm density; Testosterone; Hypogonadism
MeSH Terms: conditions — Infertility; Hypogonadism | interventions — Enclomiphene; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1(IP) (Experimental): Enclomiphene citrate capsules 25 mg 1x daily for 16 weeks
  Interventions: Drug: Enclomiphene citrate
- Arm 2 (Placebo) (Placebo Comparator): Placebo capsule 1x daily for 16 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Enclomiphene citrate — 25 mg daily for 16 weeks
  Other Names: Androxal
  Arms: Arm 1(IP)
Other: Placebo — placebo daily for 16 weeks
  Other Names: sugar pill
  Arms: Arm 2 (Placebo)

SUMMARY:
This is an exploratory, single center, randomized, parallel, double-blind placebo- and active-controlled trial in adult males ages 18 to 35 years of age who have male infertility of unknown cause. Approximately 50 men will be randomly assigned to one of two treatment groups according to a 1:1 ratio. About half of the men will receive 25mg Androxal and half of the men will receive a placebo (non-active pill) for 16 weeks. This study will last approximately 4 months and involve up to 7 visits.

The purpose of this study is to determine the effect the Androxal on sperm production.

DETAILED DESCRIPTION:
It has been estimated that 4 to 5 million men in the United States are testosterone deficient, but fewer than 10% currently receive testosterone replacement therapy. There are many reasons for the low number of men receiving testosterone replacement therapy, one of which is the route of administration. The currently approved androgen therapies are oral products, injectables, patches, buccal systems, and gels, and each has disadvantages. Oral preparations may be associated with hepatotoxicity and produce unfavorable effects on serum lipid profiles and carbohydrate metabolism. Injectables are associated with uneven levels of serum testosterone leading to fluctuations in mood, libido, and energy levels. Patches may require intrusive preparation, cause skin irritation or not adhere properly. A testosterone gel has overcome some of the above problems and has gained acceptance, but there are indications that men do not apply the gel correctly.

Previous studies showed that Androxal significantly increases total testosterone levels in men with low values at baseline. Additional studies found not only was Androxal non inferior to a topical gel, it was found to maintain sperm counts in the normal range.

Subjects will be randomized into one of the two treatment arms, using a block size of 4. The order in which the treatments are assigned in each block is randomized and this process is repeated for consecutive blocks of subjects until all subjects are randomized. This process ensures that after every fourth randomized subject, the number of subjects in each treatment group is equal.

To allow subjects in screening once the target 50 subjects have been enrolled and to account for dropouts, 75 randomization codes will be generated. As subjects are enrolled in the study, they will be assigned unique consecutive numbers starting at 001. At least 50 subjects who meet all the entry criteria will be randomized 1:1 such that approximately 25 subjects are assigned to the Androxal treatment arm and approximately 25 subjects are assigned to the placebo arm.

Placebo controlled studies are the gold standard of clinical trials and should be attempted whenever the indication and current medical practice will allow. This study is investigating a product to increase sperm concentration in subjects with idiopathic male infertility and secondary hypogonadism, low testosterone. Subjects with idiopathic male infertility do not require treatment to be healthy and approximately 18 weeks on a placebo is unlikely to harm the subjects in any way. Standard of care for idiopathic male infertility today allows subjects and physicians the option to not medically treat the disease. Therefore, the use of a placebo control in this study is well justified and will provide the best mechanism to assess treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* Men having idiopathic male infertility with sperm concentration <15million/ml (on 2 baseline semen analyses)
* Serum total testosterone < 300ng/dL if oligospermia (sperm concentration <15million/ml)
* Any testosterone if nonobstructive azoospermia (no sperm in the ejaculate)
* Men aged 18-35 living in stable relationship and desiring fertility
* Normal female partner evaluation as reported by the patient
* Ability to complete the study in compliance with the protocol
* Ability to understand and provide written informed consent

Exclusion Criteria:

* Men desiring operation for fertility (i.e. varicocelectomy) or couples desiring assisted reproductive technologies such as intrauterine insemination IUI, in vitro fertilization IVF and intracytoplasmic sperm injection ICSI) within study completion (5 months)
* Clinically significant medical condition rendering the subjects infertile including tumors of the pituitary, laboratory abnormalities
* Patients having received an investigational drug / clomiphene citrate, antioxidants, multi-vitamin in the past 30 days prior to study
* Previous treatment with androgens, estrogens, DHEA, testosterone or testosterone analogues in injectable, oral, topical or other forms for the treatment of AIHH who have not discontinued for at least 1 month prior to the start of the treatment phase
* Clinically significant abnormal findings on screening examination as determined by the investigator
* Known hypersensitivity to clomiphene citrate
* Current or history of breast cancer
* Any condition which in the opinion of the investigator would interfere with the participant's ability to provide informed consent, comply with the study instructions, possibly confound interpretation of the study results, or endanger the participant if he took part in the study
* Have received a diagnosis of irreversible infertility or compromised fertility (cryptorchidism, Kallman Syndrome, vasectomy, or tumors of the pituitary)
* Current or history of prostate cancer or a suspicion of prostate disease
* Presence or history of known hyperprolactinemia (prolactin > 17ng/dl) with or without a tumor
* Chronic use of medications use such as glucocorticoids (chronic use of inhaled or topical glucocorticoids is acceptable)
* No current drug abuse or chronic narcotic use including methadone
* Subjects with known history of HIV and/or Hepatitis C
* Subjects with end stage renal disease
* Subjects with cystic fibrosis (mutation of the CFTR gene)
* History of liver disease (including malignancy) or a confirmed AST or ALT >3 times the upper limit of normal
* History of myocardial infarction, unstable angina, symptomatic heart failure, ventricular dysrhythmia or known history of QTc interval prolongation
* History of cerebrovascular disease
* History of venous thromboembolic disease (e.g. deep vein thrombosis or pulmonary embolism)
* History of erythrocytosis or polycythemia (HCt > 54)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09-22; Primary Completion 2016-08-02 (Actual); Study Completion 2016-08-02 (Actual)

PRIMARY OUTCOMES:
Doubling of total motile sperm count | 16 weeks

SECONDARY OUTCOMES:
Morning hormone levels | 16 weeks
  Assess changes in values from baseline of total morning testosterone, estrogen and dihydrotestosterone levels after 16 weeks of treatment with placebo or 25 mg Androxal
Changes in questionnaire responses | 16 weeks
  Assess change from baseline to endpoint in Androgen Deficiency Aging Male (ADAM), International Prostate Symptom Score (I-PSS), Sexual health inventory in Male (SHIM) and psychosexual daily questionnaire (PDQ)
BMI | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Larry I. Lipshultz, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No